CLINICAL TRIAL: NCT00400205
Title: Phase II Study of Induction Docetaxel, Cisplatin and 5-Fluorouracil Chemotherapy in Squamous Cell Carcinoma of the Oral Cavity With Molecular Endpoints
Brief Title: Study of Induction Docetaxel, Cisplatin and 5-Fluorouracil
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety reasons
Sponsor: Emory University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Nabil F. Saba, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0414-2006
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Results first posted 2011-01-04 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Squamous Cell Carcinoma; Oral Cancer
Keywords: Squamous Cell Carcinoma of the Oral Cavity
MeSH Terms: conditions — Carcinoma, Squamous Cell; Mouth Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Recipients of Docetaxel, Cisplatin, 5-Fluorouracil (Experimental): Participants with squamous cell carcinoma receiving chemotherapy with docetaxel, cisplatinum, and 5-fluorouracil.
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75 mg/m2, intravenous infusion over 1 hour, mixed with normal saline per institutional standard, day 1 and then every 3 weeks.
  Other Names: Taxotere
Drug: Cisplatin — Cisplatin 100 mg/m2, intravenous infusion over 30 minutes to 3 hours, day 1 and then every 3 weeks.
Drug: 5-fluorouracil — 5-fluorouracil 1000 mg/m2/day, 24 hour continuous infusion over 4 days, every 3 weeks.

SUMMARY:
This is a Phase II study designed to test the efficacy of chemotherapy with docetaxel, cisplatinum (cisplatin) and 5-fluorouracil in patients with squamous cell carcinoma of the oral cavity to determine what effects these agents may have on cancer cells.

DETAILED DESCRIPTION:
This is a Phase II study designed to test the efficacy of chemotherapy with docetaxel, cisplatinum, and 5-fluorouracil in patients with squamous cell carcinoma of the oral cavity to determine what effects these agents may have on cancer cells.

Approximately 60 patients will take part at multi-sites with potentially 20 patients participating at the Emory Winship Cancer Institute in Atlanta, Georgia.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven squamous cell carcinoma of the oral cavity.
* Primary tumor sites eligible: oral cavity. Although they are admittedly of squamous cell types, the following tumors will be excluded because their responsiveness to chemotherapy may differ: tumors of the nasal and paranasal cavities and of the nasopharynx. Oral cavity tumors with mandible invasion are excluded because the tumor biology and management of these tumors is more complex and will likely include upfront surgical resection.
* Stage 3 or 4 disease without evidence of distant metastases verified by chest x-ray, abdominal ultrasound, or CT scan (liver function test abnormalities); bone scan in case of local symptoms.
* At least one uni- or bi-dimensionally measurable lesion.
* Age ≥ 18 years.
* World Health Organization (WHO) performance status of 2 or less.
* No active alcohol addiction.
* Final eligibility for a clinical trial is determined by the health professionals conducting the trial.

Exclusion Criteria:

* Pregnant or breast feeding
* Previous malignancies at other sites, with the exception of adequately treated in situ carcinoma of the cervix uteri, basal, or squamous cell carcinoma of the skin or other cancer curatively treated by surgery and with no evidence of disease for at least 5 years.
* Any prior treatment with radiotherapy or chemotherapy is an exclusion criterion.
* Patients who experience an involuntary weight loss of more than 25% of their body weight in the 2 months preceding study entry.
* Concurrent treatment with any other anti-cancer therapy.
* Participation in an investigational trial within 30 days of study entry.
* Patients with a history of severe hypersensitivity reaction to Taxotere® or other drugs formulated with polysorbate 80.
* No previous chemotherapy or radiotherapy for any reason and no previous surgery for SCCHN [squamous cell carcinoma of the head and neck] (other than biopsy) are allowed at the time of study entry.
* Final eligibility for a clinical trial is determined by the health professionals conducting the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Saba, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Result] Saba NF, Magliocca KR, Kim S, Muller S, Chen Z, Owonikoko TK, Sarlis NJ, Eggers C, Phelan V, Grist WJ, Chen AY, Ramalingam SS, Chen ZG, Beitler JJ, Shin DM, Khuri FR, Marcus AI. Acetylated tubulin (AT) as a prognostic marker in squamous cell carcinoma of the head and neck. Head Neck Pathol. 2014 Mar;8(1):66-72. doi: 10.1007/s12105-013-0476-6. Epub 2013 Jul 24. PMID 23881549

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Accrual period is from Aug 2006 through Jul 2009. Accrual of 14 patients.
Pre-assignment Details: A total of 14 patients with squamous carcinoma were enrolled. All patients had stage 4a or 4b disease and had a performance status of 0-2 then all had measurable lesions on imaging. The study closed prematurely due to slow accrual and increased observed complications.
Groups:
- Recipients of Docetaxel, Cisplatin, 5-Fluorouracil: Participants with squamous cell carcinoma receiving chemotherapy with docetaxel, cisplatin, and 5-fluorouracil
Period: Overall Study
Arm/Group | Recipients of Docetaxel, Cisplatin, 5-Fluorouracil
Started | 14
Completed | 9
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- Recipients of Docetaxel, Cisplatin, 5-Fluorouracil: Patients with locally advanced squamous cell carcinoma of the head and neck received three cycles of induction therapy with docetaxel, cisplatin, and 5-fluorouracil followed by local therapy consisting of surgical resection in addition to possible radiation therapy with or without concurrent chemotherapy.
Arm/Group | Recipients of Docetaxel, Cisplatin, 5-Fluorouracil
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 14
Tumor Stage IV [Number; unit: Participants] — Cancer stage was assessed with the tumor, node and metastasis (TNM) staging system. The TNM Classification of Malignant Tumors is a commonly used system of assessing cancer severity. Stage IV refers to cancer that has spread to distant body parts and is the most severe stage.
  Participants | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Had Response by RECIST Criteria (Response Evaluation Criteria in Solid Tumors)
Description: Complete remission (complete disappearance of disease), partial remission [more than 30% decrease in tumor measurement by RECIST (Response evaluation criteria in solid tumors)].
Time Frame: every 3 months
Measure: Number; unit: participants
Arm/Group | Recipients of Docetaxel, Cisplatin, 5-Fluorouracil
Number analyzed (Participants) | 9
participants | 8

2. Secondary Outcome: Tumor Change by Baseline Acetylated Tubulin Expression Score
Description: Percent change in TNM stage of tumors after three cycles of study treatment was assessed to see if baseline acetylated tubulin (AT) expression predicts treatment success. Decreasing tumor stage change (a negative number) indicates that the tumor is responding to treatment while an increase means that the severity of the tumor is not decreasing. Immunohistochemistry (IHC) analysis of AT expression was performed in formalin-fixed, paraffin-embedded, pre-treatment tissues. The staining was scored based upon intensity according to the following criteria: 0=no staining, 1+=weak tumor staining, 2+=moderate tumor staining, 3+=moderate to high tumor staining, and 4+=high tumor staining.
  Data presented are adopted from Saba, NF, et. al. Acetylated Tubulin (AT) as a Prognostic Marker in Squamous Cell Carcinoma of the Head and Neck. Head and Neck Pathology (2014) 8:66-72.
Time Frame: Baseline, After 3 cycles of study treatment
Population: Participants who completed the study are included in this analysis.
Measure: Mean (Standard Deviation); unit: percentage of tumor stage change
Arm/Group | Recipients of Docetaxel, Cisplatin, 5-Fluorouracil
Number analyzed (Participants) | 9
percentage of tumor stage change
  AT score less than or equal to 2: number analyzed (Participants) | 4
  AT score less than or equal to 2 | -0.8 (0.23)
  AT score greater than 2: number analyzed (Participants) | 5
  AT score greater than 2 | -0.36 (0.44)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Recipients of Docetaxel, Cisplatin, 5-Fluorouracil
All-Cause Mortality (participants affected / at risk) | 3/14
Serious Adverse Events (participants affected / at risk) | 6/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recipients of Docetaxel, Cisplatin, 5-Fluorouracil (N=14)
Death (Infections and infestations) | 1 (1)
Death (General disorders) | 1 (1)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Fever neutropenia (Infections and infestations) | 1 (1)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PEG tube infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recipients of Docetaxel, Cisplatin, 5-Fluorouracil (N=14)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 7 (8)
Cellulitis (Skin and subcutaneous tissue disorders) | 7 (9)
Constipation (Gastrointestinal disorders) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Dehydration (Metabolism and nutrition disorders) | 7 (7)
Depression (Psychiatric disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 6 (9)
Difficulty speaking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dizziness (General disorders) | 6 (12)
Dry mouth (General disorders) | 4 (4)
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Facial pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Fatigue (General disorders) | 12 (23)
Fever (General disorders) | 6 (11)
Heartburn (Gastrointestinal disorders) | 3 (3)
Hypokalemia (Blood and lymphatic system disorders) | 6 (7)
Insomnia (General disorders) | 11 (12)
Loss of appetite (General disorders) | 9 (10)
Mouth pain (General disorders) | 12 (37)
Mucositis (Gastrointestinal disorders) | 10 (21)
Nausea (General disorders) | 9 (13)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (9)
Neuropathy (Nervous system disorders) | 4 (4)
Odynophagia (Gastrointestinal disorders) | 5 (15)
Oral thrush (Infections and infestations) | 7 (7)
Restlessness (Nervous system disorders) | 3 (3)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Vision disturbance (Eye disorders) | 2 (2)
Vomiting (General disorders) | 5 (5)
Weakness (General disorders) | 7 (8)
Weight loss (General disorders) | 9 (16)
Mouth sores (Gastrointestinal disorders) | 5 (5)
Edema (Metabolism and nutrition disorders) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes